CLINICAL TRIAL: NCT02683642
Title: Invasive Mould Infections in Indian ICUs - Descriptive Epidemiology, Management and Outcome
Status: Completed | Type: Observational
Sponsor: Fungal Infection Study Forum (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Arunaloke Chakrabarti, Chairman, FISF, Fungal Infection Study Forum
Other Study IDs: FungalISF
Record Dates: First submitted 2015-12-21; First posted 2016-02-17 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Mycoses
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Invasive mould infections are emerging causes of morbidity and mortality in ICU patients. This is attributed to prolonged ICU stay of critically ill patients with many co-morbidities. Modern medicine and multiple intervention make the patients susceptible to these prevalent moulds in the environment. In India the high frequency of IMIs in general has been attributed to environmental and host factors prevalent in this region. Additionally sub-optimal hospital care practice, frequent demolition and construction activities in the hospital make the patients susceptible to IMIs. There is no multicentric study available in India describing the epidemiology of IMIs in India. However, single center studies have reported distinct epidemiology of IMIs in India. High incidence, different spectrum and risk factors are possible unique features of IMIs in India.Early diagnosis and optimal therapy improve the outcome of these patients. The conventional diagnosis including histopathology and culture has limitations. The tests are of low sensitivity and long turnaround time. The major challenge is collection of sample from deep tissue. Therefore majority of the patients in ICUs of India are managed empirically against invasive fungal diseases. The galactomannan test has improved the diagnosis of invasive aspergillosis. However, galactomannan test is not well standardized in non-neutropenic patients. Beta-glucan test is used for early diagnosis of invasive fungal infections other than mucormycosis. But the test is cumbersome for routine laboratories and expensive. Both tests are not available in majority of Institutions of India. PCR assay is not standardized and not performed routinely in any Institution.

Due these limitations in diagnosis, there is no uniform management protocol in ICUs of India. To develop optimal management protocol, we need to know the epidemiology, the right patient to treat, antifungal drug resistance, optimal drug and duration of therapy etc. The present study will provide descriptive epidemiology, present status of diagnosis and management practiced in India to treat IMIs in ICUs. This will help to find the suitable intervention strategies to improve outcome of IMIs in India.This descriptive observational prospective study will document the epidemiologic and clinical characteristics, as well as treatment and outcome data, of patients with IMIs in ICUs in India over one year.

DETAILED DESCRIPTION:
The prospective study will describe the epidemiology of IMIs in ICUs in India. The study will describe the incidence, risk factors, fungi causing IMIs and their susceptibility against antifungal agents, as well as the current strategies adopted by ICU physicians in the management of IMIs. It will also describe the outcome of IMIs. The study will help in planning future management strategies specific for IMIs in ICUs in India.

Methods

Study description: Prospective, multicenter study in iCUs in India.

Purpose: Determination of epidemiologic parameters, including risk factors, description of current management and outcome of patients with IMI will be recorded prospectively. The study will help in understanding the epidemiology of IMI in ICUs and possible planning for future management strategies for IMI specific to India.

Risk: There is no risk to the patient from the study as it is only an observational study and no intervention is intended.

Site selection: 15 ICU's are identified across the country where ICU physicians are well versed about invasive fungal infections and competent diagnostic mycology laboratory is available

A site feasibility survey was conducted. This ensured that participating sites fulfill the following inclusion criteria: a) maintains ICD coding and total number of discharges and deaths at the center; b) manages critically ill patients in ICU; c) has access to high-resolution CT (HRCT) scans; d) has a mycology laboratory that performs isolation and identification of fungi at least perform galactomannan test; and e) has histopathology facilities.

Study Period: April 1, 2016 to June 30, 2017. Case enrolment - April 1, 2016 to March 31, 2017. Analysis of data - April 1, 2017 to June 30, 2017

No. of patients: All consecutive patients with proven and probable IMI in ICUs at the study centers during the study period will be included.

Patient selection All consecutive patients diagnosed for proven or probable IMIs in ICUs at the study sites will be included.

Inclusion criteria:

Proven:

Histopathology/cytology/culture/direct microscopy demonstrating septate hyphae invading tissue or aspirate from sterile sites

Probable:

* Host satisfies host criteria of EORTC
* Host with COPD satisfying definitions by Bulpa P, et al Eur Resp J 2007
* Host in ICU satisfying clinical algorithm by Blot SI, et al Am J Resp Crit Care Med 2012

Exclusion criteria:

* Endemic mycoses (histoplasmosis, sporotrichosis, penicilliosis)
* Yeast infections
* Allergic fungal diseases like allergic bronchopulmonary aspergillosis
* Infection limited to the skin only

Conduct of the study

Investigators of the study: Arunaloke Chakrabarti will be the coordinator of the study. Each site will have a Principal Investigator - the site PI. Other investigators at the site will be co-investigators.

Patient enrollment: The site PI (or one of the co-investigators) will review the patient's paper and electronic records to determine if the patient satisfies the inclusion criteria. Patients who fulfill the inclusion criteria will be included as a case.

Data collection: The demographic, clinical, treatment and outcome data will be collected by investigator and email the form to the study coordinator, Arunaloke Chakrabarti. Outcome will be measured on day of discharge/death/30 and 120 days (whichever is earlier) after the diagnosis of the IMI. The date of diagnosis of an IMI is the day on which the diagnosis is defined as proven or probable. For cases that were enrolled as probable but subsequently became proven, the date of diagnosis is the earlier date. In addition, each center will also obtain data from its relevant hospital authority on the total number of discharges and deaths in ICUs for the period of April 1, 2016 to March 31, 2017.

Fungal isolates: All isolates from proven and probable IMIs will be sent to Mycology Reference Laboratory at PGIMER, Chandigarh for final identification and antifungal susceptibility testing

Patient management: The study will not interfere with patient management.

Statistics

The study will be analyzed using descriptive statistics. It is anticipated that the study will provide the following information:

* Incidence of IMI among patients in ICUs during the study period in the participating centers
* Relative frequency of each risk factor among IMI patients at the participating centers.
* Three-month survival of patients diagnosed with IMI.
* Other data the study should be able to generate will be in accordance with the objectives.
* Kaplan-Meier plots will be used to describe the survival of patients with IMI according to their underlying diagnosis.

ELIGIBILITY:
Inclusion criteria:

Proven:

Histopathology/cytology/culture/direct microscopy demonstrating septate hyphae invading tissue or aspirate from sterile sites

Probable:

* Host criteria of EORTC
* Host with COPD satisfying definitions by Bulpa P, et al Eur Resp J 2007
* Host in ICU satisfying clinical algorithm by Blot SI, et al Am J Resp Crit Care Med 2012

Exclusion criteria:

* Endemic mycoses (histoplasmosis, sporotrichosis, penicilliosis)
* Yeast infections
* Allergic fungal diseases like allergic bronchopulmonary aspergillosis
* Infection limited to the skin only

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 15 ICU are identified across the country where ICU physicians are well versed about invasive fungal infections and competent diagnostic mycology laboratory is available
  A site feasibility survey was conducted. This ensured that participating sites fulfill the following inclusion criteria: a) maintains ICD coding and total number of discharges and deaths at the center; b) manages critically ill patients in ICU; c) has access to high-resolution CT (HRCT) scans; d) has a mycology laboratory that performs isolation and identification of fungi at least perform galactomannan test; and e) has histopathology facilities.
  All consecutive patients with proven and probable IMI in ICUs at the study centers during the study period will be included.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Invasive mould infections (IMIs) in Indian ICUs (Number of patients with IMI per 1000 ICU admissions) | Three months from the date of admission

SECONDARY OUTCOMES:
Incidence in specific population (Number of patients with IMI in specific population per 1000 ICU admissions) | six months after the completion of the study
Mortality (number of deaths per 1000 ICU admissions) | six months after the completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Arunaloke Chakrabarti, MD, DNB, Study Director — PGIMER, Chandigarh; Shivaprakash M Rudramurthy, MD, Principal Investigator — PGIMER, Chandigarh; Randeep Guleria, MD, Principal Investigator — AIIMS, New Delhi; Malini Capoor, MD, Principal Investigator — Vardhman Mahavir Medical College, New Delhi; Arvind Baronia, MD, Principal Investigator — SGPGI, Lucknow; Subhash Todi, MD, Principal Investigator — AMRI Hospitals, Kolkata; Sanjay Bhattacharyya, MD, Principal Investigator — Tata Medical Centre, Kolkata; P Umabala, MD, Principal Investigator — NIMS, Hyderabad; Ranganathan Iyer, MD, Principal Investigator — Global Hospital, Hyderabad; Ram Gopalakrishnan, MD, Principal Investigator — Apollo Hspital, Chennai; Anupma J Kindo, MD, Principal Investigator — Sri Ramchandra Medical University, Chennai; O C Abraham, MD, Principal Investigator — CMC, Vellore; Sriram Sampath, MD, Principal Investigator — St John Medical College, Bengaluru; Rajeev Soman, MD, Principal Investigator — Hinduja Hospital, Mumbai; Atul Patel, MD, Principal Investigator — Sterling Hospital, Ahmedabad; Pradip Bhattacharyya, MD, Principal Investigator — Chirayu Medical College, Bhopal
Locations (11):
- India (11):
  - Sterling Hospital, Ahmedabad, Gujarat
  - St.Johns Medical College, Bangalore, Karnataka
  - Chirayu Medical College, Bhopal, Madhya Pradeh
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Sri Ramchandra Medical university, Chennai, Tamil Nadu
  - Christian Medical College, Vellore, Tamil Nadu
  - Nizams Institute Of Medical Sciences, Hyderabad, Telangana
  - AMRI Hospital, Kolkata, West Bengal
  - PGIMER, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chakrabarti A, Kaur H, Savio J, Rudramurthy SM, Patel A, Shastri P, Pamidimukkala U, Karthik R, Bhattacharya S, Kindo AJ, Bhattacharya P, Todi S, Gopalakrishan R, Singh P, Pandey A, Agarwal R. Epidemiology and clinical outcomes of invasive mould infections in Indian intensive care units (FISF study). J Crit Care. 2019 Jun;51:64-70. doi: 10.1016/j.jcrc.2019.02.005. Epub 2019 Feb 5. PMID 30769292